CLINICAL TRIAL: NCT01062399
Title: Phase I/II Trial of Concurrent RAD001 (Everolimus) With Temozolomide/Radiation Followed by Adjuvant RAD001/Temozolomide in Newly Diagnosed Glioblastoma
Brief Title: Everolimus, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Acronym: RTOG 0913
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0913; RTOG-0913; CDR0000664302; NCI-2011-00885 (Registry Identifier: CTRP: (Clinical Trials Reporting Office))
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Everolimus; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Ph I: RT + TMZ + RAD001 2.5 mg/day (Experimental): Radiation therapy (RT), concurrent temozolomide (TMZ), and concurrent RAD001 2.5 mg/day followed by post-radiation temozolomide and post-radiation RAD001 10 mg/day.
  Interventions: Drug: concurrent temozolomide; Radiation: Radiation therapy; Drug: concurrent RAD001 2.5 mg/day; Drug: post-radiation RAD001 10 mg/day; Drug: post-radiation temozolomide
- Ph I: RT + TMZ + RAD001 5 mg/day (Experimental): Radiation therapy, concurrent temozolomide, and concurrent RAD001 5 mg/day followed by post-radiation temozolomide and post-radiation RAD001 10 mg/day.
  Interventions: Drug: concurrent temozolomide; Radiation: Radiation therapy; Drug: concurrent RAD001 5 mg/day; Drug: post-radiation RAD001 10 mg/day; Drug: post-radiation temozolomide
- Ph I: RT + TMZ + RAD001 10 mg/day (Experimental): Radiation therapy, concurrent temozolomide, and concurrent RAD001 10 mg/day followed by post-radiation temozolomide and post-radiation RAD001 10 mg/day.
  Interventions: Drug: concurrent RAD001 10 mg/day; Drug: concurrent temozolomide; Radiation: Radiation therapy; Drug: post-radiation RAD001 10 mg/day; Drug: post-radiation temozolomide
- Ph II: RT + TMZ (Active Comparator): Radiation therapy and concurrent temozolomide followed by post-radiation temozolomide
  Interventions: Drug: concurrent temozolomide; Radiation: Radiation therapy; Drug: post-radiation RAD001 10 mg/day; Drug: post-radiation temozolomide
- Ph II: RT + TMZ + RAD001 (Experimental): Radiation therapy, concurrent temozolomide, and concurrent RAD001 10 mg/day followed by post-radiation temozolomide and post-radiation RAD001 10 mg/day.
  Interventions: Drug: concurrent RAD001 10 mg/day; Drug: concurrent temozolomide; Radiation: Radiation therapy; Drug: post-radiation RAD001 10 mg/day; Drug: post-radiation temozolomide

INTERVENTIONS:
Drug: concurrent RAD001 10 mg/day — During radiation: RAD001 10 mg orally daily during radiation therapy; one hour prior to radiation and in the morning on weekends on days 1-42.
  Other Names: everolimus
  Arms: Ph I: RT + TMZ + RAD001 10 mg/day; Ph II: RT + TMZ + RAD001
Drug: concurrent temozolomide — During radiation: temozolomide 75 mg/m2/day orally daily during radiation therapy; one hour prior to radiation and in the morning on weekends on days 1-42. Dose rounded to the nearest 5 mg.
Radiation: Radiation therapy — Intensity Modulated RT (IMRT) allowed. For both IMRT and 3D conformal radiotherapy (3D-CRT) plans, one treatment of 2 Gy given daily 5 days per week for a total of 60 Gy over 6 weeks.
Drug: concurrent RAD001 2.5 mg/day — During radiation: RAD001 2.5 mg orally daily during radiation therapy; one hour prior to radiation and in the morning on weekends on days 1-42.
  Other Names: everolimus
  Arms: Ph I: RT + TMZ + RAD001 2.5 mg/day
Drug: concurrent RAD001 5 mg/day — During radiation: RAD001 5 mg orally daily during radiation therapy; one hour prior to radiation and in the morning on weekends on days 1-42.
  Other Names: everolimus
  Arms: Ph I: RT + TMZ + RAD001 5 mg/day
Drug: post-radiation RAD001 10 mg/day — Post-radiation: RAD001 10 mg orally daily on days 1-28 of each cycle, for up to 12 cycles, starting 28 days after the completion of radiation therapy (Cycle = 28 days).
  Other Names: everolimus
Drug: post-radiation temozolomide — Post-radiation: temozolomide 150 mg/m2/day - 200 mg/m2/day orally daily on days 1-5 of each cycle, starting 28 days after the completion of radiation therapy for up to 12 cycles (Cycle = 28 days)

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells. Giving everolimus together with temozolomide and radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of everolimus when given together with temozolomide and radiation therapy and to see how well it works in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define the maximum tolerated dose of everolimus (up to an established dose of 10 mg/day) when combined with concurrent radiotherapy and temozolomide in patients with newly diagnosed glioblastoma multiforme. (Phase I)
* To determine the efficacy of everolimus in combination with radiotherapy and temozolomide followed by adjuvant everolimus in combination with temozolomide, as measured by progression-free survival, in these patients. (Phase II)

Secondary

* To characterize the safety profile of everolimus in combination with radiotherapy and temozolomide in these patients. (Phase I)
* To determine the overall survival of these patients. (Phase II)
* To further evaluate the safety profile of everolimus in combination with radiotherapy and temozolomide in these patients. (Phase II)
* To determine if activation of the Akt/mTOR axis predicts response to everolimus. (Phase II)
* To determine if there is an association between tumor MGMT gene methylation status and response to everolimus. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of everolimus followed by a phase II, randomized study.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion criteria:

1. Histologically proven diagnosis of glioblastoma (WHO grade IV) confirmed by central pathology review prior to Step 2 registration. Since gliosarcoma is a variant of glioblastoma, gliosarcoma is also an eligible diagnosis.
2. Tumor tissue available for correlative studies (Required only in phase II portion, as described below).

   * Patients must have at least 1 block of tissue; if a block cannot be submitted, two tissue specimens punched with a skin punch (2 mm diameter) from the tissue block containing the tumor may be submitted.
   * Diagnosis must be made by surgical excision, either partial or complete. Stereotactic biopsy or Cavitron ultrasonic aspirator (CUSA)-derived tissue is not allowed for patients on Phase II, as it will not provide sufficient tissue for the required MGMT and pAKT/pMTOR analyses.
3. The tumor must have a supratentorial component
4. Patients must have recovered from the effects of surgery, postoperative infection, and other complications.
5. A diagnostic contrast-enhanced MRI or CT scan (if MRI is not available due to non-compatible devices) of the brain must be performed preoperatively and postoperatively. The postoperative scan must be done within 28 days prior to step 2 registration, ,preferably within 96 hours of surgery. Preoperative and postoperative scans must be the same type.

   • Patients unable to undergo MRI imaging because of non-compatible devices can be enrolled, provided pre- and post-operative contrast enhanced CT scans are obtained and are of sufficient quality.
6. History/physical examination within 14 days prior to step 2 registration
7. Neurologic examination within 14 days prior to step 2 registration
8. Documentation of steroid doses within 14 days prior to step 2 registration
9. Karnofsky performance status ≥ 70
10. Age ≥ 18 years
11. Complete blood count (CBC)/differential obtained within 14 days prior to step 2 registration, with adequate bone marrow function defined as follows:

    * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3;
    * Platelets ≥ 100,000 cells/mm3;
    * Hemoglobin ≥ 10.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is acceptable.)
12. Prothrombin time/international normalized ratio (PT INR) ≤ 1.5 for patients not on warfarin confirmed by testing within 14 days prior to step 2 registration.

    Patients on full-dose anticoagulants (eg, warfarin or low molecular weight heparin) must meet both of the following criteria:
    * No active bleeding or pathological condition that carries a high risk of bleeding (eg, tumor involving major vessels or known varices)
    * In-range INR (between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
13. Adequate renal function, as defined below:

    * Blood urea nitrogen (BUN) ≤ 30 mg/dl within 14 days prior to step 2 registration
    * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) within 14 days prior to step 2 registration
14. Adequate hepatic function, as defined below:

    * Bilirubin ≤ 1.5 x normal range within 14 days prior to step 2 registration
    * Alanine aminotransferase (ALT) ≤ 2.5 x normal range within 14 days prior to step 2 registration
    * Aspartate aminotransferase (AST) ≤ 2.5 x normal range within 14 days prior to step 2 registration
15. Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN (upper limit of normal). Note: If one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
16. For females of child-bearing potential, negative serum pregnancy test within 14 days prior to step 2 registration
17. Women of childbearing potential and male participants must practice adequate contraception
18. Patient must provide study-specific informed consent prior to registration

Exclusion criteria:

1. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
2. Recurrent or multifocal malignant glioma
3. Metastases detected below the tentorium or beyond the cranial vault
4. Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment
5. Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation therapy fields
6. Prior chemotherapy or radiosensitizers for cancer of the head and neck region; note that prior chemotherapy for a different cancer is allowable, except prior temozolomide or RAD001.
7. Prior radiation therapy or chemotherapy for glioblastoma
8. Severe, active co-morbidity, defined as follows:

   * Symptomatic congestive heart failure of New York heart Association Class III or IV
   * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within the last 6 months, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
   * Severely impaired lung function as defined as spirometry and diffusing capacity of the lungs for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
   * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
   * Active (acute or chronic) or uncontrolled severe infections requiring intravenous antibiotics
   * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
   * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition or known HIV seropositivity; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with HIV/AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity
   * Other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2010-12; Primary Completion 2016-06 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Chinnaiyan, MD, Principal Investigator — William Beaumont Hospital and Oakland University School of Medicine
Locations (36):
- United States (34):
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - St. Vincent Oncology Center, Indianapolis, Indiana
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario, Canada
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Result] Chinnaiyan P, Won M, Wen PY, Rojiani AM, Wendland M, Dipetrillo TA, Corn BW, Mehta MP. RTOG 0913: a phase 1 study of daily everolimus (RAD001) in combination with radiation therapy and temozolomide in patients with newly diagnosed glioblastoma. Int J Radiat Oncol Biol Phys. 2013 Aug 1;86(5):880-4. doi: 10.1016/j.ijrobp.2013.04.036. Epub 2013 May 29. PMID 23725999
- [Result] Chinnaiyan P, Won M, Wen PY, Rojiani AM, Werner-Wasik M, Shih HA, Ashby LS, Michael Yu HH, Stieber VW, Malone SC, Fiveash JB, Mohile NA, Ahluwalia MS, Wendland MM, Stella PJ, Kee AY, Mehta MP. A randomized phase II study of everolimus in combination with chemoradiation in newly diagnosed glioblastoma: results of NRG Oncology RTOG 0913. Neuro Oncol. 2018 Apr 9;20(5):666-673. doi: 10.1093/neuonc/nox209. PMID 29126203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 279 patients registered at 1st registration for central pathology review of histology confirmation. Among 279 patients, 72 patients did not go beyond 2nd step registration due to insufficient tissue, patient refusal, progression of disease, and other reasons.
Period: Overall Study
Arm/Group | Ph I: RT + TMZ + RAD001 2.5 mg/Day | Ph I: RT + TMZ + RAD001 5 mg/Day | Ph I: RT + TMZ + RAD001 10 mg/Day | Ph II: RT + TMZ | Ph II: RT + TMZ + RAD001
Started | 8 | 10 | 8 | 89 | 92
Completed | 8 (Subjects with data available for the primary analyses are considered to have completed the study.) | 9 | 8 | 83 | 88
Not Completed | 0 | 1 | 0 | 6 | 4
Not completed — Protocol Violation | 0 | 1 | 0 | 6 | 4

BASELINE CHARACTERISTICS:
Population: Eligible randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph I: RT + TMZ + RAD001 2.5 mg/Day | Ph I: RT + TMZ + RAD001 5 mg/Day | Ph I: RT + TMZ + RAD001 10 mg/Day | Ph II: RT + TMZ | Ph II: RT + TMZ + RAD001 | Total
Number analyzed (Participants) | 8 | 9 | 8 | 83 | 88 | 196
Age, Continuous [Median (Full Range); unit: years] | 58 [39 to 72] | 57 [39 to 69] | 57 [31 to 73] | 57 [23 to 79] | 61 [25 to 82] | 59 [23 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 6 | 37 | 32 | 80
  Male | 4 | 8 | 2 | 46 | 56 | 116

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Patients With Dose-limiting Toxicity (DLT)
Description: DLT is defined as any of the following events occurring during the first 8 weeks of treatment with RAD001 and temozolomide and attributable to the study drugs: any grade 3 or 4 thrombocytopenia, grade 4 anemia, or grade 4 neutropenia lasting more than 7 days; any non-hematologic grade 3 or greater adverse event (AE), excluding alopecia, despite maximal medical therapy; any grade 4 radiation-induced skin changes; failure to recover from adverse events to be eligible for re-treatment with RAD001 and temozolomide within 14 days of the last dose of either drug; or any episode of non-infectious pneumonitis grade 2, 3, or 4 of any duration. Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE
Time Frame: From start of treatment to eight weeks.
Population: First 6 eligible phase I patients at each dose level who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ph I: RT + TMZ + RAD001 2.5 mg/Day | Ph I: RT + TMZ + RAD001 5 mg/Day | Ph I: RT + TMZ + RAD001 10 mg/Day
Number analyzed (Participants) | 6 | 6 | 6
Participants | 2 | 2 | 2
Statistical Analysis 1: Comparison: Ph I: RT + TMZ + RAD001 2.5 mg/Day vs Ph I: RT + TMZ + RAD001 5 mg/Day vs Ph I: RT + TMZ + RAD001 10 mg/Day; Test type: Other; A dose level for RAD001 will be considered acceptable if no patient of the first 3patients or no more than 2 patients of the first 6 patients experience a DLT. If the current level is considered acceptable, then dose escalation will occur and the protocol will be reopened. Otherwise, the preceding acceptable dose level will be declared the MTD

2. Primary Outcome: Phase II: Progression-free Survival (PFS)
Description: Using the Response Assessment in Neuro- Oncology (RANO) criteria, the progression is defined by any of the following: > 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared to the smallest tumor measurement obtained either at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids; Significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation of therapy, not due to co-morbid events; Any new lesion; Clear clinical deterioration not attributable to other causes apart from the tumor or changes in corticosteroid dose; Failure to return for evaluation due to death or deteriorating condition; Clear progression of non-measurable disease. PFS time is defined as time from registration to date of progression, death, or last known follow-up (censored). PFS rates are estimated using the Kaplan-Meier method.
Time Frame: Analysis occured after 134 events (progression or death) were reported. Patients were followed from randomization to death or study termination whichever occurs first, up to 36.7 months.
Population: Eligible phase II patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ph II: RT + TMZ | Ph II: RT + TMZ + RAD001
Number analyzed (Participants) | 83 | 88
months | 10.2 [7.5 to 13.8] | 8.2 [6.5 to 10.6]
Statistical Analysis 1: Comparison: Ph II: RT + TMZ vs Ph II: RT + TMZ + RAD001; Assuming exponential distribution with median PFS (mPFS) time for control of 6.7 mos. for the control arm, tt was hypothesized that there would be a 43% improvement in mPFS time, corresponding to a mPFS time of 9.6. This is equivalent to a hazard ratio of 0.7 for the experimental arm vs. control arm. With a 1-sided significance level = 0.15 and 85% power, a total of 134 PFS events out of 180 eligible patients were required to detect the projected effect size; Test type: Superiority; p = 0.79, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.82 to 1.60] — Reference arm = RT + TMZ

3. Secondary Outcome: Phase II: Overall Survival (OS)
Description: Overall survival time is defined as time from/randomization to the date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: as for outcome 2
Population: Eligible phase II patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ph II: RT + TMZ | Ph II: RT + TMZ + RAD001
Number analyzed (Participants) | 83 | 88
months | 21.2 [16.6 to 29.9] | 16.5 [12.5 to 18.7]
Statistical Analysis 1: Comparison: Ph II: RT + TMZ vs Ph II: RT + TMZ + RAD001; Test type: Superiority; p = 0.008, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 1.67, 95% CI 2-sided [1.14 to 2.45] — Reference level = RT + TMZ

4. Secondary Outcome: Phase I: Distribution of Worst Adverse Event Grade
Description: AE reporting in Phase I was split up by treatment timing: concurrent treatment (RT, TMZ, RAD001); post-RT treatment (TMZ, RAD001) along with all AE's reported in follow-up.
  The worst/highest grade of any adverse event reported in each time period was determined for each patient. The percentage of patients in each grade level is reported. Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: as for outcome 2
Population: Eligible phase I patients who started the corresponding study treatment and had adverse events assessed.
Measure: Number; unit: percentage of participants
Arm/Group | Ph I: RT + TMZ + RAD001 2.5 mg/Day | Ph I: RT + TMZ + RAD001 5 mg/Day | Ph I: RT + TMZ + RAD001 10 mg/Day
Number analyzed (Participants) | 8 | 9 | 8
percentage of participants
  Concurrent treatment: Grade 1 | 0.0 | 11.1 | 12.5
  Concurrent treatment: Grade 2 | 0.0 | 33.3 | 0.0
  Concurrent treatment: Grade 3 | 50.0 | 44.4 | 87.5
  Concurrent treatment: Grade 4 | 50.0 | 11.1 | 0.0
  Concurrent treatment: Grade 5 | 0.0 | 0.0 | 0.0
  Post-RT treatment: Grade 1: number analyzed (Participants) | 7 | 7 | 3
  Post-RT treatment: Grade 1 | 0.0 | 0.0 | 0.0
  Post-RT treatment: Grade 2: number analyzed (Participants) | 7 | 7 | 3
  Post-RT treatment: Grade 2 | 0.0 | 42.9 | 100.0
  Post-RT treatment: Grade 3: number analyzed (Participants) | 7 | 7 | 3
  Post-RT treatment: Grade 3 | 71.4 | 28.6 | 0.0
  Post-RT treatment: Grade 4: number analyzed (Participants) | 7 | 7 | 3
  Post-RT treatment: Grade 4 | 14.3 | 0.0 | 0.0
  Post-RT treatment: Grade 5: number analyzed (Participants) | 7 | 7 | 3
  Post-RT treatment: Grade 5 | 14.3 | 0.0 | 0.0

5. Secondary Outcome: Phase II: Distribution of Worst Adverse Event Grade
Description: The worst/highest grade of any adverse event reported was determined for each patient. The percentage of patients in each grade level is reported. Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: as for outcome 2
Population: Eligible phase II patients who started study treatment and had adverse events assessed.
Measure: Number; unit: percentage of patients
Arm/Group | Ph II: RT + TMZ | Ph II: RT + TMZ + RAD001
Number analyzed (Participants) | 77 | 85
percentage of patients
  Grade 1 | 0 | 0
  Grade 2 | 0 | 3
  Grade 3 | 3 | 5
  Grade 4 | 3 | 0
  Grade 5 | 2 | 1

ADVERSE EVENTS:
Description: Eligible patients who started study treatment and had adverse events assessed are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Ph I: RT + TMZ + RAD001 2.5 mg/Day | Ph I: RT + TMZ + RAD001 5 mg/Day | Ph I: RT + TMZ + RAD001 10 mg/Day | Ph II: RT + TMZ | Ph II: RT + TMZ + RAD001
Serious Adverse Events (participants affected / at risk) | 6/8 | 3/9 | 2/8 | 17/77 | 49/85
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 8/8 | 76/77 | 85/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ph I: RT + TMZ + RAD001 2.5 mg/Day (N=8) | Ph I: RT + TMZ + RAD001 5 mg/Day (N=9) | Ph I: RT + TMZ + RAD001 10 mg/Day (N=8) | Ph II: RT + TMZ (N=77) | Ph II: RT + TMZ + RAD001 (N=85)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 3
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Death NOS (General disorders) | 1 | 1 | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 6
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Cranial nerve infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Duodenal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Scrotal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 1 | 0 | 1 | 10
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 5
Platelet count decreased (Investigations) | 1 | 1 | 0 | 2 | 11
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 1 | 0 | 0 | 1 | 8
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Edema cerebral (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 3 | 9
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 2 | 0 | 0 | 1 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Thromboembolic event (Vascular disorders) | 2 | 0 | 0 | 2 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ph I: RT + TMZ + RAD001 2.5 mg/Day (N=8) | Ph I: RT + TMZ + RAD001 5 mg/Day (N=9) | Ph I: RT + TMZ + RAD001 10 mg/Day (N=8) | Ph II: RT + TMZ (N=77) | Ph II: RT + TMZ + RAD001 (N=85)
Anemia (Blood and lymphatic system disorders) | 6 | 3 | 6 | 24 | 53
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1 | 5
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 2 | 2 | 5
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 1 | 8 | 10
Cushingoid (Endocrine disorders) | 2 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 2 | 1 | 2 | 9 | 13
Dry eye (Eye disorders) | 1 | 0 | 0 | 2 | 0
Optic nerve disorder (Eye disorders) | 1 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 3
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 2 | 4 | 38 | 36
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 2 | 13 | 16
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 7
Mucositis oral (Gastrointestinal disorders) | 3 | 4 | 3 | 6 | 32
Nausea (Gastrointestinal disorders) | 4 | 5 | 5 | 42 | 48
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 15 | 22
Edema limbs (General disorders) | 1 | 1 | 1 | 10 | 16
Fatigue (General disorders) | 8 | 4 | 7 | 67 | 68
Fever (General disorders) | 2 | 1 | 1 | 7 | 9
Gait disturbance (General disorders) | 2 | 0 | 0 | 7 | 5
Irritability (General disorders) | 2 | 0 | 0 | 2 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 0 | 0 | 2 | 2
Mucosal infection (Infections and infestations) | 3 | 0 | 1 | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 0 | 0 | 2 | 6
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 25 | 27
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 3
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 4
Alanine aminotransferase increased (Investigations) | 4 | 4 | 4 | 28 | 41
Aspartate aminotransferase increased (Investigations) | 5 | 4 | 5 | 19 | 38
Blood bilirubin increased (Investigations) | 3 | 1 | 0 | 9 | 10
CD4 lymphocytes decreased (Investigations) | 4 | 2 | 3 | 11 | 8
Cholesterol high (Investigations) | 8 | 6 | 8 | 21 | 56
Creatinine increased (Investigations) | 3 | 0 | 1 | 6 | 17
INR increased (Investigations) | 1 | 0 | 0 | 0 | 4
Investigations - Other (Investigations) | 2 | 0 | 1 | 6 | 12
Lymphocyte count decreased (Investigations) | 7 | 7 | 8 | 43 | 49
Neutrophil count decreased (Investigations) | 2 | 3 | 6 | 19 | 27
Platelet count decreased (Investigations) | 7 | 4 | 6 | 37 | 55
Weight loss (Investigations) | 3 | 1 | 4 | 7 | 18
White blood cell decreased (Investigations) | 5 | 4 | 7 | 36 | 45
Anorexia (Metabolism and nutrition disorders) | 5 | 4 | 3 | 25 | 34
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 3 | 3 | 30 | 44
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 8 | 4
Hypernatremia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 1 | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6 | 6 | 6 | 14 | 53
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 2 | 0 | 7 | 17
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 12 | 23
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1 | 2 | 7 | 23
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 11 | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6 | 12
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 15 | 13
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 4 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 4
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 4
Ataxia (Nervous system disorders) | 1 | 1 | 2 | 6 | 9
Cognitive disturbance (Nervous system disorders) | 2 | 0 | 0 | 10 | 11
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 7 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 2 | 18 | 12
Dysgeusia (Nervous system disorders) | 2 | 1 | 4 | 16 | 25
Headache (Nervous system disorders) | 6 | 5 | 7 | 41 | 40
Memory impairment (Nervous system disorders) | 3 | 2 | 0 | 26 | 13
Nervous system disorders - Other (Nervous system disorders) | 1 | 0 | 1 | 14 | 6
Paresthesia (Nervous system disorders) | 1 | 2 | 1 | 2 | 3
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 2 | 3 | 0 | 15 | 16
Tremor (Nervous system disorders) | 2 | 0 | 0 | 6 | 7
Agitation (Psychiatric disorders) | 4 | 1 | 0 | 4 | 5
Anxiety (Psychiatric disorders) | 2 | 0 | 1 | 13 | 11
Confusion (Psychiatric disorders) | 3 | 2 | 1 | 10 | 12
Depression (Psychiatric disorders) | 4 | 0 | 0 | 15 | 11
Insomnia (Psychiatric disorders) | 4 | 1 | 1 | 19 | 17
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 0 | 4 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 4 | 4
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 5 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 2 | 7 | 44 | 49
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 7 | 8
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 7 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 5 | 8
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 4 | 12
Scalp pain (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 4 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 7 | 7
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 3
Hypotension (Vascular disorders) | 1 | 0 | 1 | 3 | 7
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 4 | 6
Vascular disorders - Other (Vascular disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.